CLINICAL TRIAL: NCT04584229
Title: Chemsex Among Men Who Have Sex With Men : Perceived Risks and Coping Strategies, a Qualitative Study.
Brief Title: Chemsex, Perceived Risks and Coping Strategies.
Acronym: Chemsex
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0091
Record Dates: First submitted 2020-10-06; First posted 2020-10-12 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Sexual; Sexual Desire; Illicit Drugs; MSM
Keywords: screening; MSM; Qualitative research; HIV transmission; men who have sex with men; Risk Reduction Behavior; Harm Reduction; recreational drugs; Sexualised drug use
MeSH Terms: conditions — Coitus; Substance-Related Disorders; Homosexuality; Risk Reduction Behavior; Harm Reduction | interventions — Methods

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- question not suitable for study: question not suitable for study
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — Intervention: comprehensive individual or collective interview, recorded and transcribed

SUMMARY:
The research hypothesis is that access to prevention and harm and risk reduction associated with the use of psychoactive substances in a sexual context is insufficient for MSM practicing chemsex. This would lead to a lack of awareness of the risks taken and insufficient or inadequate strategies to protect themselves.

This qualitative study has a comprehensive objective. The aim is to identify the risks perceived by MSM practicing Chemsex and their coping strategies. The study is based on individual semi-directed interviews and focus group. The criteria for inclusion are: an age greater than or equal to 18 years, being a man having sex with men and having used psychoactive substances in a sexual context at least once in the past 12 months. Participants were recruited through a gay geo-social networking app on mobile phones on a voluntary basis. At the same tim+e, flyers presenting the study are also distributed to the "chemsex" consultations at the Montpellier University Hospital in France as well as to an association fighting against AIDS in Montpellier.

Data are subjected to an inductive method analysis, bringing out by constant comparison conceptualizing categories illustrating the experience and making it possible to identify and understand the risks felt and the coping strategies.

ELIGIBILITY:
Inclusion criteria:

* an age greater than or equal to 18 years
* being a man having sex with men
* having used psychoactive substances in a sexual context at least once in the past 12 months.

Exclusion criteria:

- to refuse to participate to the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men who have sex with other men
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Chemsex Paretic Risk Assessment | 1 day
  Chemsex Paretic Risk Assessment

SECONDARY OUTCOMES:
Description of the population leaving Chemsex | 1 day
  Description of the population leaving Chemsex

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Donnadieu-Rigole, MD, PHD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC